CLINICAL TRIAL: NCT04756869
Title: Monitoring Health Care Workers at Risk for COVID-19 Using Wearable Sensors and Smartphone Technology
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Sung Won Choi, Edith S Briskin and Shirley K Schlafer Foundation Research Professor of Pediatrics and Associate Professor of Pediatrics and Communicable Diseases, University of Michigan
Other Study IDs: HUM00180076
Record Dates: First submitted 2021-02-15; First posted 2021-02-16 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Covid19
Keywords: mobile health; wearable sensors; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Subjects will provide self-collected nasal and saliva samples up to daily during the study period. These samples will be used to test for SARS-CoV-2, which will help to establish an estimate of the asymptomatic carrier frequency in the health care worker population. Subjects can also opt-in to providing blood samples at up to three time points within a year of enrollment, with a goal of determining baseline and changes in antibody titers to SARS-CoV-2, as well as obtaining specimens for the measurement of other immunologic parameters and biomarkers - including immune cell profiling and DNA/RNA-seq analysis. Subjects that receive a diagnosis of COVID-19 while on-study may provide additional nasal swabs, saliva, and/or blood specimens up to 1 year after study completion.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Health Care Workers at Risk for COVID-19: Health care workers at risk for COVID-19 will be monitored using wearing sensors and smartphone technology.
  Interventions: Other: COVID-19 Monitoring Using Wearable Sensors and Smartphone Technology

INTERVENTIONS:
Other: COVID-19 Monitoring Using Wearable Sensors and Smartphone Technology — Health care workers are on-study for 30 days, in which they wear a smart watch and temperature patches up to daily. Subjects also may provide nasal and saliva samples up to daily during the study period, and they may opt-in to blood samples lasting up to 1 year after study completion. Through a smartphone app, participants complete surveys at baseline and at study completion, as well as daily mood surveys and symptom-reporting surveys. Finally, exit interviews occur at the end of the study period, and follow-up interviews may occur at specified timepoints up to 1 year after study completion.

SUMMARY:
This prospective study of health care workers utilizes wearable sensors, surveys and symptom logs, and biospecimens in an effort to improve self-monitoring practices for COVID-19 among health care workers and to provide key data for the development of a predictive model for early detection of COVID-19 infection.

DETAILED DESCRIPTION:
Health care workers work on the front lines of the COVID-19 pandemic, so early detection of COVID-19 infection is especially important in this population in order to prevent the spread of disease among the health care workforce, their patients, and their families. However, standard symptomatic COVID-19 testing is insufficient to protect health care workers and prevent the spread of disease. This study utilizes continuous physiological data from wearable sensors and surveys completed via smartphone technology, in conjunction with biospecimens, in order to assist health care workers in their self-monitoring for COVID-19 infection. Subjects will wear smart watches and temperature monitoring patches to collect continuous heart rate and temperature data. Subjects will also complete baseline and exit surveys, in addition to daily mood and symptom logging surveys. Finally, subjects will provide biospecimens - nasal and saliva samples and optional blood samples. Using wearable sensor data in conjunction with survey data and biospecimens, this study aims to prevent the spread of COVID-19 among health care workers, their patients, and their families, and to eventually develop a predictive model for early detection of COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* Adult Michigan Medicine health care workers age 18 years and older.
* Health care workers who are involved in direct (in-person) face-to-face patient care or health care workers who are not involved in direct (in-person) face-to-face patient care but work on units where COVID-19 patients are/will likely be treated.
* Possession of a smartphone (Apple or Android).
* Ability to understand and demonstrate willingness to remotely sign a written informed consent.

Exclusion Criteria:

* Unwilling or unable to comply with the study procedures or to allow the study team access to health data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health care workers at Michigan Medicine at risk for COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2021-01-16 (Actual); Study Completion 2021-01-16 (Actual)

PRIMARY OUTCOMES:
Feasibility of Wearing Fitbit Watch | 30 days
  Feasibility is defined as wearing the Fitbit Watch for at least 8 hours a day, 5 days a week (~40 hours/week or 160 hours/30 days).
Feasibility of Wearing TempTraq Patch | 30 days
  Feasibility is defined as wearing the TempTraq for at least 8 hours a day, five days a week (~40 hours/week or 160 hours/30 days).

SECONDARY OUTCOMES:
Survey Completion Rate | 30 days
  This outcome is measured by the percentage of subjects that complete their surveys, estimating that at least 50% of subjects will complete the baseline and exit surveys, and at least 50% of subjects will complete at least 50% of the daily symptom surveys.

OTHER OUTCOMES:
Clinical Health Outcomes | 2 years
  Detection of SARS-CoV-2 using any of the following: biospecimens, self-reported test results, a database of COVID-19 testing and results maintained in Employee Health at Michigan Medicine, and subjects' electronic medical records

CONTACTS AND LOCATIONS:
Overall Officials: Sung Choi, MD, MS, Principal Investigator — University of Michigan
Locations (1):
- Michigan Medicine, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be shared with other researchers when the appropriate Data Use Agreement (DUA) is in place. What IPD will be shared is undecided at this time.

REFERENCES:
- [Derived] Clingan CA, Dittakavi M, Rozwadowski M, Gilley KN, Cislo CR, Barabas J, Sandford E, Olesnavich M, Flora C, Tyler J, Mayer C, Stoneman E, Braun T, Forger DB, Tewari M, Choi SW. Monitoring Health Care Workers at Risk for COVID-19 Using Wearable Sensors and Smartphone Technology: Protocol for an Observational mHealth Study. JMIR Res Protoc. 2021 May 12;10(5):e29562. doi: 10.2196/29562. PMID 33945497